CLINICAL TRIAL: NCT02402907
Title: A Randomized Trial to Determine if a Pre-operative Wash With a Chlorhexidine Cloth Reduces Infectious Morbidity in Patients Undergoing Cesarean Section
Brief Title: STRIPES Study: Study To Reduce Infection Post cEsarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne L Stone, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GCO 14-1410
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Chlorhexidine Gluconate Cloths; Infection; Cesarean Section; Infectious Morbidity; Surgical Site Infections; Endometritis
Keywords: cesarean section; chlorhexidine gluconate; CHG; surgical site infection; obstetrics; infection prevention; pregnancy
MeSH Terms: conditions — Infections; Surgical Wound Infection; Endometritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHG cloth (Experimental): 2% chlorhexidine gluconate (CHG) cloth
  Interventions: Device: 2% chlorhexidine gluconate (CHG) cloth
- Placebo cloth (Placebo Comparator): A fragrance free cleansing cloth
  Interventions: Device: Placebo cloth

INTERVENTIONS:
Device: 2% chlorhexidine gluconate (CHG) cloth — administration of a 2% CHG cloth at home on the night before and approximately 3 hours prior to cesarean delivery on the morning of the surgery.
  Other Names: CHG
  Arms: CHG cloth
Device: Placebo cloth — administration of a cloth with the placebo (commercial cleansing cloth) at home on the night before and approximately 3 hours prior to cesarean delivery on the morning of the surgery.
  Other Names: Cleansing cloth
  Arms: Placebo cloth

SUMMARY:
The objective of this study is to determine if the use of chlorhexidine gluconate cloths prior to cesarean section reduce the rate of infectious morbidity (i.e. surgical site infections, endometritis).

The study will be offered to women who present for a scheduled primary or repeat cesarean section at Mount Sinai Medical Center. The eligible women will be randomized to use of a 2% chlorhexidine gluconate (CHG) cloth or placebo cloth (a fragrance free cleansing cloth) the night before and the morning of their scheduled procedure. Participants will be blinded to the arm in which they have been assigned. This study intends to show that the use of 2% CHG cloths prior to cesarean section will reduce the rate of surgical site infections.

DETAILED DESCRIPTION:
Chlorhexidine is a sterile, germ-free solution, which is regularly used to clean the skin immediately before surgery and works by killing or preventing the growth or spread of bacteria. Data exists in both the orthopedic and cardiac literature to show that an additional preoperative use of chlorhexidine further reduces the risk of post procedure infections. Limited data exists regarding the use of a preoperative use of chlorhexidine in patients undergoing Obstetric or Gynecologic procedures and there is no wash or cloth used prior to cesarean section as a standard of care. The hope for this study is to identify if an additional preoperative chlorhexidine wash will further decrease or prevent infection in women who deliver their babies via cesarean section.

All patients with a scheduled cesarean section surgery will be approached for enrollment during their pre-admission testing visit on the labor floor 2 days before the scheduled cesarean section, a visit that is standard procedure for this surgery. Once a patient is consented, she will be randomly assigned to one of the 2 arms of the study: the eligible women will be randomized to use of 2% chlorhexidine gluconate (CHG) cloths or placebo cloths (a fragrance free cleansing cloths) on the body the night before and the morning of their scheduled procedure. Participants will be blinded to the arm in which they have been assigned.

The purpose of this study is to determine if the use of 2% chlorhexidine gluconate cloths prior to cesarean section reduces the rate of surgical site wound infection and/or postpartum endometritis, which is an infection or inflammation of the endometrium (the inner lining of the uterus).

ELIGIBILITY:
Inclusion Criteria:

* women
* > 24 weeks gestation
* scheduled for a primary or repeat cesarean section

Exclusion criteria:

* allergy to chlorhexidine
* unplanned or emergency cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1356 (Actual)
Dates: Start 2015-04; Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Stone, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1356 were enrolled, 14 did not undergo procedure at Sinai, leaving 1342 participants (672 in experimental group and 670 in placebo group) that continued on the study.
Groups:
- Placebo Cloth: Placebo cloth: administration of a fragrance free cleansing cloth with the placebo (commercial cleansing cloth) at home on the night before and approximately 3 hours prior to cesarean delivery on the morning of the surgery.
Period: Overall Study
Arm/Group | CHG Cloth | Placebo Cloth
Started | 682 | 674
Completed | 662 | 647
Not Completed | 20 | 27
Not completed — Delivered vaginally | 9 | 3
Not completed — Delivered outside of Sinai | 1 | 1
Not completed — Lost to follow up after C-Section | 10 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHG Cloth | Placebo Cloth | Total
Number analyzed (Participants) | 682 | 674 | 1356
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age
  years | 35.1 (5.0) | 35.1 (5.0) | 35.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 682 | 674 | 1356
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 66 | 60 | 126
  White | 436 | 416 | 852
  Hispanic or Latino | 113 | 121 | 234
  Unknown or Not Reported | 67 | 77 | 144
Private Insurance [Count of Participants; unit: Participants] | 604 | 577 | 1181
Chronic Hypertension [Count of Participants; unit: Participants] | 23 | 26 | 49
Pregestational Diabetes [Count of Participants; unit: Participants] | 9 | 13 | 22
Asthma [Count of Participants; unit: Participants] | 47 | 28 | 75
Primiparous [Count of Participants; unit: Participants] | 248 | 236 | 484
Repeat Cesarean Delivery [Count of Participants; unit: Participants] | 387 | 394 | 781
Gestational Hypertension [Count of Participants; unit: Participants] | 17 | 18 | 35
Gestational Diabetes [Count of Participants; unit: Participants] | 69 | 57 | 126
Preeclampsia [Count of Participants; unit: Participants] | 8 | 13 | 21
Cholestasis [Count of Participants; unit: Participants] | 8 | 7 | 15
Estimated Blood loss [Median (Inter-Quartile Range); unit: mL] — Population: Data results only for those participants who underwent C-Section at Sinai
  mL
    number analyzed (Participants) | 672 | 670 | 1342
    (all) | 719.5 [479.5 to 800.0] | 717.5 [484.0 to 800] | 718.5 [479.5 to 800]
Length of procedure [Median (Inter-Quartile Range); unit: min] — Population: Data results only for those participants who underwent C-Section at Sinai
  min
    number analyzed (Participants) | 672 | 670 | 1342
    (all) | 62.0 [53.0 to 74.0] | 62.0 [53.0 to 76.0] | 62.0 [53.0 to 76.0]
Preincision Prophylactic Antibiotics [Count of Participants; unit: Participants] — Population: Data results only for those participants who underwent C-Section at Sinai
  Participants
    Clindamycin/gentamicin: number analyzed (Participants) | 672 | 670 | 1342
    Clindamycin/gentamicin | 14 | 12 | 26
    Cefazolin | 645 | 648 | 1293
Skin Closure Type [Count of Participants; unit: Participants] — Population: Data results only for those participants who underwent C-Section at Sinai
  Participants
    Staples: number analyzed (Participants) | 672 | 670 | 1342
    Staples | 56 | 58 | 114
    Subcuticular suture | 616 | 612 | 1228

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incisional SSI
Description: Number of participants with Incisional Surgical Site Infection (SSI)
Time Frame: at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 662 | 647
Participants | 17 | 24

2. Primary Outcome: Number of Adherent Participants With Incisional SSI
Description: Among those with full adherence to the protocol and who were available for assessment at 6 weeks. Adherence to the protocol was assessed in the following 2 ways: evaluation of returned packages on the day of surgery and report ascertained by phone interview at 2 weeks.
Time Frame: at 6 weeks
Population: participants with full adherence to protocol and available for assessment at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 524 | 515
Participants | 10 | 17

3. Primary Outcome: Number of Participants With Endometritis
Description: Number of participants with endometritis
Time Frame: at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 662 | 647
Participants | 0 | 1

4. Secondary Outcome: Number of Participants With Maternal Complications
Description: Number of participants with maternal complications
Time Frame: up to 6 weeks
Population: Data results only for those participants who underwent C-Section at Sinai
Measure: Count of Participants; unit: Participants
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 672 | 670
Participants
  Erythema at operative site | 16 | 16
  Skin Separation | 19 | 23
  Drainage | 21 | 16
  Fever | 4 | 2
  Hematoma | 1 | 5
  Seroma | 2 | 0

5. Secondary Outcome: Incidence of Neonatal ICU Admissions
Time Frame: up to 6 weeks
Population: Data not collected
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Maternal Length of Stay
Description: Length of stay (index hospitalization)
Time Frame: at 6 weeks
Population: data for participants who were hospitalized
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 652 | 651
days | 3.0 [3.0 to 3.0] | 3.0 [3.0 to 3.0]

7. Secondary Outcome: Number of Participants With Maternal Readmissions
Description: Number of participants with hospital readmission for wound complication
Time Frame: up to 6 weeks
Population: Data results only for those participants who underwent C-Section at Sinai. unable to obtain data for 2 participants in placebo cloth arm
Measure: Count of Participants; unit: Participants
Arm/Group | CHG Cloth | Placebo Cloth
Number analyzed (Participants) | 672 | 668
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | CHG Cloth | Placebo Cloth
All-Cause Mortality (participants affected / at risk) | 0/672 | 0/670
Serious Adverse Events (participants affected / at risk) | 0/672 | 0/670
Other Adverse Events (participants affected / at risk) | 0/672 | 0/670

LIMITATIONS AND CAVEATS:
Limitations included the lower than anticipated rate of SSIs after scheduled cesarean deliveries, suggesting the possibility that the study was underpowered for the primary outcome. High rate of private insurance may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT02402907/Prot_SAP_000.pdf